CLINICAL TRIAL: NCT00391235
Title: White Matter Connectivity in Pediatric Bipolar Disorder: A Diffusion Tensor Imaging Study
Brief Title: White Matter in Pediatric Bipolar Disorder: A DTI Study
Status: Completed | Type: Observational
Sponsor: Cambridge Health Alliance (Other)
Collaborators: American Academy of Child Adolescent Psychiatry. (Other); Eli Lilly and Company (Industry)
Responsible Party: Jean Frazier, MD, Cambridge Health Alliance
Other Study IDs: CHA-IRB-0132/09/05
Record Dates: First submitted 2006-10-19; First posted 2006-10-23 (Estimated); Last update posted 2010-12-06 (Estimated); Status verified 2010-12

CONDITIONS: Bipolar Disorder
Keywords: bipolar disorder; magnetic resonance imaging; white matter; diffusion tensor imaging; children; adolescents
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- BPD: Children with bipolar disorder
- HC: Healthy comparison children

SUMMARY:
Fourteen subjects with bipolar disorder and 14 matching healthy controls, aged 6-13, will receive a magnetic resonance imaging (MRI) scan on a 3 Tesla scanner. They will also have a clinical interview, including the KSADS-PL. All subjects must be right-handed.

DETAILED DESCRIPTION:
We propose to investigate the connectivity of white matter tracts using diffusion tensor imaging (DTI) in children with very early onset bipolar disorder (BPD). We hypothesize that the connectivity between the prefrontal cortex and the temporal lobe and parietal lobe and limbic structures will be abnormal, indicating white matter and gray matter deficits in early onset BPD. We also hypothesize that the superior lateral fasciculus cingulum bundle and the inferior lateral fasciculus will have decreased fractional anisotropy in very early onset BPD relative to healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 to 13
* Male or female
* Right-handed

Exclusion Criteria:

* IQ less than 70
* Learning disabilities
* History of autism, schizophrenia, anorexia or bulimia nervosa
* Substance abuse
* Claustrophobia
* Metal in body
* Pregnancy or lactation

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Bipolar Disorder
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2005-09; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Fractional anisotropy in brain white matter | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jean A Frazier, MD, Principal Investigator — Cambridge Health Alliance
Locations (1):
- Cambridge Health Alliance, Medford, Massachusetts, United States

REFERENCES:
- See also: Description of this research program at Cambridge Health Alliance — http://www.cha.harvard.edu/ccad/index.shtml